CLINICAL TRIAL: NCT05164224
Title: Correlation of Serum Procalcitonin and Severity of Post-cesarean Wound Infection
Brief Title: Serum Procalcitonin and Post-cesarean Wound Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Elsibai Anter, Assistant professor of obstetrics and gynecology, Menoufia University
Other Study IDs: 12/2020 BSGN 14
Record Dates: First submitted 2021-12-05; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Cesarean Wound Disruption

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No secondary suture: The participants who will develop post-cesarean surgical site infection and follow-up only antibiotic treatment for their wound care.
- secondary suture: The participants who will develop post-cesarean surgical site infection and need a secondary suture for their wound care

SUMMARY:
serum procalcitonin levels are important during infections and sepsis.The aim of this study is to evaluate the correlation between serum procalcitonin and severity of post cesarean wound infection

DETAILED DESCRIPTION:
Bacterial infection is primarily a clinical concept that may require the use of supportive bedside or laboratory tests to confirm or exclude. There are two broad factors that are always necessary to confirm the diagnosis: inflammation or systemic dysfunction and direct or indirect evidence of a compatible bacterial pathogen. Inflammation may be localized or result in a systemic inflammatory response syndrome (SIRS).

Infection handling and prevention are now improving with an effective antibiotic discovery, complete immunization and modern sanitation. However, infection remains the most common cause of morbidity and mortality rate in many health care services in the world.

One of the most often serious complications in surgical procedure is surgical site infection. Surgical site infection (SSI) is defined as the presence of liquid pus or abscess which extends on a wound within 30day (RCOG Press, 2008; Bratzlr et al.,2006). Surgical site infection is diagnosed with clinical and laboratory examination. The diagnosis begins with an inspection to check any pus, abscess or inflammation reaction extends on the surgical site. An open wound is also being checked, as well as pus liquid or abscess that leaks from thewound. Pus or tissue specimen should be taken for culture examination and routine blood count for leucocyte count should be investigated and procalcitonin level Procalcitonin (PCT) and leucocyte count are indicators of systemic infection. Procalcitonin is one of the applicable markers to detect bacterial infection in adults. Plasma PCT level is comparable with specific response of bacterial infection, particularly for invasive or probably-invasive bacteria. High concentration of PCT indicates sepsis, severe sepsis or even septic shock condition. It may also represent another possibility and gives additional information towards conventional clinical data. Some studies state that procalcitonin is better, or at least has the same diagnosis potency with another infection marker such as CRP, leukocytosis and fever

ELIGIBILITY:
Inclusion Criteria:

* patients who will develop surgical site infection after their cesarean sections.
* 18-40 years old

Exclusion Criteria:

* History of chorioamnionitis, premature rupture of membranes or prolonged rupture of membrane.
* Urinary tract infections.
* Any infectious condition other than surgical site infection.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Patients planned for cesarean section
Study Population: patients who will develop surgical site infection after their cesarean sections
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Serum procalcitonin levels in participants who will developwound infection after cesarean sections | 2 weeks
  Serum procalcitonin levels will be measured in participants who will develop post-cesarean wound site infections. The serum procalcitonin levels will be compared in subgroups (who need secondary suture and those who willn't require suturing)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Anter, MD, Study Director — Menoufia University-Shebin Elkom-Egypt
Locations (1):
- Menoufia University hospital, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes